CLINICAL TRIAL: NCT04537429
Title: An Open-label, Single-dose, Pharmacokinetic Study to Evaluate IV Eptinezumab in Children and Adolescents With Migraine, Followed by an Optional, Multiple-dose, Open-label Extension Period
Brief Title: A Study in Children and Young People With Migraine to Learn What the Body Does to Eptinezumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18922A
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Migraine in Children; Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eptinezumab (Experimental)
  Interventions: Drug: Eptinezumab

INTERVENTIONS:
Drug: Eptinezumab — up to four iv infusions of eptinezumab

SUMMARY:
The purpose of the study is to investigate how the body absorbs, distributes, and get rid of eptinezumab when given directly into a vein.

DETAILED DESCRIPTION:
This is an interventional, open-label pharmacokinetic study with eptinezumab, consisting of a single-dose, 20-week main study period (Part A) and an optional 44-week multiple-dose extension period (Part B).

The main study period includes a single IV infusion of eptinezumab. The optional extension period includes 3 additional eptinezumab infusions 12 weeks apart (reflecting recommended dosing interval in adults), for a total of up to 4 infusions over the course of the study.

At least 32 patients with migraine will be enrolled: 16 patients aged 6 to 11 years, and 16 patients aged 12 to 17 years, inclusive.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of migraine with or without aura according to international classification of headache disorders (ICHD)-3 (in the opinion of the investigator) for ≥6 months prior to the Screening Visit and has a frequency of migraine ≥4 migraine days per month for at least 3 months prior to the Screening Visit.

Exclusion Criteria:

* The patient has been exposed to any monoclonal antibody treatment (including exposure in a study) <6 months prior to the Screening Visit.

Other in- and exclusion criteria may apply

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) (0-infinity) eptinezumab | From dosing to week 20
  Area under the plasma concentration curve for eptinezumab from zero to infinity
Cmax eptinezumab | From dosing to week 20
  Maximum observed plasma concentration of eptinezumab

SECONDARY OUTCOMES:
Clearance (CL) | From dosing to week 20
  Plasma clearance
Volume of distribution (Vz) | From dosing to week 20
Development of anti-eptinezumab antibodies (ADA) | From screening to week 12
Characterization of anti-eptinezumab antibodies for neutralizing activity (NAb) | From screening to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (9):
- United States (9):
  - New England Institute for Clinical Research, Stamford, Connecticut
  - NW FL Clinical Research Group LLC, Gulf Breeze, Florida
  - The Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - College Park Family Care Center, Overland Park, Kansas
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Preferred Primary Care Physicians Inc., Pittsburgh, Pennsylvania
  - North Texas Institute of Neurology & Headache, Frisco, Texas
  - Road Runner Research Ltd, San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah